CLINICAL TRIAL: NCT05460273
Title: Phase 1/2, Multicentre, Open-label, Multiple-cohort Study of Dato-DXd in Chinese Patients With Advanced Non-small-cell Lung Cancer, Triple-negative Breast Cancer, Gastric/Gastroesophageal Junction Cancer, Urothelial Cancer, and Other Solid Tumours (TROPION-PanTumor02)
Brief Title: A Study of Dato-DXd in Chinese Patients With Advanced Non-Small Cell Lung Cancer, Triple-negative Breast Cancer and Other Solid Tumors (TROPION-PanTumor02)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9266C00001
Record Dates: First submitted 2022-06-08; First posted 2022-07-15 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Cancer
Keywords: Non-small-cell Lung Cancer; Triple-negative Breast Cancer; Dato-DXd; DS-1062a
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/Phase 2, multicentre, open-label, multiple-cohort study, which is designed to evaluate the efficacy, safety, PK, and immunogenicity of Dato-DXd in adult Chinese participants with advanced or metastatic solid tumours.
Masking Description: It is a single-arm, multi-cohort study with no blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dato-DXd Arm (Experimental): This single-arm study consists of multiple cohorts, divided by indication.
  Interventions: Drug: Datopotamab Deruxtecan (Dato-DXd)

INTERVENTIONS:
Drug: Datopotamab Deruxtecan (Dato-DXd) — Dato-DXd is an antibody-drug conjugate (ADC) that binds to TROP2.
  Other Names: DS-1062a

SUMMARY:
Researchers are looking for a better way to treat advanced Triple-Negative Breast Cancer (TNBC) and Non-Small-Cell Lung Cancer (NSCLC). "Advanced" usually means that the cancer keeps growing even with treatment. The cancer may also be "metastatic", which means that it has spread to other parts of the body or the surrounding tissue.

The study drug, Datopotamab deruxtecan, is designed to work by attaching to the tumor cells and stopping the tumor growth. Datopotamab deruxtecan is also known as Dato-DXd.

In this study, the researchers want to find out how well Dato-DXd works to stop tumors from growing in Chinese participants with NCSLC or TNBC. This is the first time Dato-DXd is being studied in Chinese population.

Participants in this study will get Dato-DXd through a needle as an injection. They will get 1 dose of Dato-DXd every 3 weeks until their cancer gets worse or they leave the study for another reason.

Participants will visit their study sites at least once every 3 weeks for as long as they are in the study. The study doctors will take blood samples every 3 weeks and take images of the participants' tumors every 6 weeks until the participant leaves the study.

DETAILED DESCRIPTION:
This is a Phase 1/Phase 2, multicentre, open-label, multiple-cohort study, which is designed to evaluate the efficacy, safety, Pharmacokinetic, and immunogenicity of Dato-DXd in adult Chinese participants with advanced or metastatic solid tumours. It is a single-arm study with no blinding.

This study is divided into different cohorts. Participants of the same cohort are with the same tumour type. The starting cohorts are Cohort 1 (NSCLC) and Cohort 2 (TNBC). Future cohorts will consist of other advanced or metastatic solid tumour types, including, but not limited to, advanced/unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma or urothelial carcinoma that is refractory or intolerant to SoC therapy or for which no Standard of Care therapy is available.

Cohort 1 and Cohort 2 will be prioritised for immediate enrolment and the protocol will be amended as needed for the future cohorts.

Cohort 1: The target population of Cohort 1 is adult Chinese participants with advanced or metastatic NSCLC with or without actionable genomic alterations(AGAs) (ie, alterations in genes with approved therapies, such as EGFR, ALK, or other known AGAs).

Eligible participants without AGAs will have been previously treated with platinum-based chemotherapy and anti-PD-1/anti-PD-L1 monoclonal antibody either in combination or sequentially. Participants without AGAs who received anti-PD-1/anti-PD-L1 monoclonal antibody as frontline therapy may have received the combination of platinum-based chemotherapy and anti-PD-1/anti-PD-L1 monoclonal antibody in the second-line setting.

Eligible participants with AGAs will have been previously treated with one or two prior lines of applicable targeted therapy that is approved for the participant's genomic alteration and platinum-based chemotherapy as the only prior line of cytotoxic therapy. Participants with AGAs may have received up to one anti-PD-1/anti-PD-L1 monoclonal antibody treatment alone or in combination with chemotherapy.

A total of approximately 40 eligible participants in China will be enrolled in this cohort, including approximately 6 participants with AGAs.

Cohort 2: The target population of Cohort 2 is adult Chinese participants with inoperable locally advanced or metastatic TNBC who have received at least 2 prior chemotherapy regimens for advanced breast cancer, counting the (neo)adjuvant therapy as a prior chemotherapy regimen if progression occurred within 12 months after completion of the therapy (DFI ≤ 12 months).

A total of approximately 78 eligible participants in China will be enrolled in this cohort. Cohort 2 will enroll at most around 20% (approximately N=15) of enrolled participants with a DFI ≤ 12 months.

Enrolled participants will be treated with Dato-DXd at 6.0 mg/kg via an IV infusion on Day 1,every 3 weeks.

The primary objective of the study is to estimate the effectiveness of Dato-DXd by assessment of confirmed ORR by independent central review.

ELIGIBILITY:
Key Inclusion Criteria:

* Capable of giving signed informed consent.
* Participant must be ≥ 18 years at the time of screening.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* At least one lesion not previously irradiated that qualifies as a RECIST 1.1 target lesion at baseline and can be accurately measured at baseline and is suitable for accurate repeated measurements.

Additional Inclusion Criteria for Cohort 1 (NSCLC):

- Histologically or cytologically documented Stage IIIB or IIIC NSCLC disease not amenable for surgical resection or definitive chemoradiation or Stage IV NSCLC disease at the beginning of study intervention.

For the subset of participants without AGAs:

* Documented negative test results for EGFR and ALK genomic alterations. If test results for EGFR and ALK are not available, participants are required to undergo testing performed locally for these genomic alterations.
* Participants must meet one of the required prior therapy requirements for advanced or metastatic NSCLC.

For the subset of participants with AGAs:

- Documented positive test results for one or more actionable genomic alteration: EGFR, ALK, ROS1, METex14 skipping, RET or other AGAs with approved therapies

- Received one or two prior lines of applicable targeted therapy for the participant's genomic alteration at the time of screening.

Additional Inclusion Criteria for Cohort 2 (TNBC)

* Pathologically documented oestrogen and progesterone receptor-negative and HER2-negative expression.
* Inoperable locally advanced or metastatic breast cancer.
* Received at least 2 prior chemotherapy regimens for locally advanced or metastatic breast cancer and previously treated with a taxane in any setting.

Key Exclusion Criteria:

* Has leptomeningeal carcinomatosis or metastasis
* Has clinically significant corneal disease
* Has known active hepatitis or uncontrolled hepatitis B or C infection
* Has a history of non-infectious ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Prior exposure to specific therapies without an adequate treatment washout period prior to enrolment.

Additional Exclusion Criteria for Cohort 1 (NSCLC):

- Has mixed SCLC and NSCLC histology.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Shenyang
  - Research Site, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9266C00001&attachmentIdentifier=40bd669c-9d78-427d-b670-1dc0ba7734e0&fileName=d9266c00001-csp-v4-Redacted_on_21Aug2024-updated.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9266C00001&attachmentIdentifier=e7e43d4e-e301-401e-8a57-641fff9615c9&fileName=d9266c00001-sap-ed-2_Redacted_on_21Aug2024.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9266C00001&attachmentIdentifier=712dc6b5-d58d-4fec-93b9-2439c4fb078d&fileName=d9266c00001-study-synopsis-NSCLC&TNBC_clean-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1/2, open-label, multiple-cohort, single-arm study was conducted in participants with Advanced Non-Small-Cell Lung Cancer (NSCLC) and Triple-Negative Breast Cancer(TNBC) in China.
  * For TNBC cohort, first participant was screened on 11Jul2022, last participant was screened on 27Apr2023.
  * For NSCLC cohort, first participant was screened on 29Aug2022, last participant was screened on 21Mar2023.
Pre-assignment Details: Overall 168 participants were screened at 23 centers in China. A total of 119 participants were treated with Dato-DXd.
  * For TNBC cohort, 106 participant was screened at 14 centers in China. 79 participants received Dato-DXd at the 14 centers.
  * For NSCLC cohort, 62 participant was screened at 12 centers in China. 40 participants received Dato-DXd at 11 centers.
  Note: 3 centers screened both TNBC participants and NSCLC participants.
Groups:
- TNBC Cohort: Final Analysis with DCO on 06May2024
- NSCLC Cohort: Primary Analysis with DCO on 09Oct2023
Period: Overall Study
Arm/Group | TNBC Cohort | NSCLC Cohort
Started | 79 | 40
Completed | 29 | 0 (NSCLC cohort has not reached final analysis.)
Not Completed | 50 | 40
Not completed — Death | 43 | 9
Not completed — Lost to Follow-up | 7 | 0
Not completed — Ongoing participants at NSCLC primary analysis DCO | 0 | 31

BASELINE CHARACTERISTICS:
Population: FAS: Enrolled participants who have received at least one dose of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | TNBC Cohort | NSCLC Cohort | Total
Number analyzed (Participants) | 79 | 40 | 119
Age, Customized [Number; unit: Participants]
  <50 | 39 | 6 | 45
  50-65 | 31 | 20 | 51
  65-75 | 9 | 14 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 11 | 90
  Male | 0 | 29 | 29
Race/Ethnicity, Customized [Number; unit: Participants]
  ASIAN | 79 | 40 | 119
Region of Enrollment [Number; unit: Participants]
  China | 79 | 40 | 119

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate(ORR) Assessed by Independent Central Review(ICR)
Description: Confirmed ORR is defined as the proportion of participants in each cohort who have a confirmed CR or confirmed PR, as assessed by ICR per RECIST 1.1.
Time Frame: TNBC cohort: from enrollment to 12 months post last subject dose with an average of 12 months follow up. NSCLC cohort: from enrollment to 6 months post last subject dose with an average of 8 months follow up.
Population: RES: Enrolled participants who received at least one dose of study intervention and had measurable disease at baseline by ICR.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 77 | 40
Percentage of participants | 33.8 [23.4 to 45.4] | 45.0 [29.3 to 61.5]

2. Secondary Outcome: Confirmed Objective Response Rate(ORR) Assessed by Investigator
Description: Confirmed ORR is defined as the proportion of participants in each cohort who have a confirmed CR or confirmed PR, as determined by investigator assessment per RECIST 1.1.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 77 | 40
Percentage of participants | 31.2 [21.1 to 42.7] | 32.5 [18.6 to 49.1]

3. Secondary Outcome: Duration of Response (DoR), Assessed by Investigator
Description: Duration of response is defined as the time from the date of first documented response (which is subsequently confirmed) until date of documented progression per RECIST 1.1, as assessed by investgator, or death due to any cause.
Time Frame: as for outcome 1
Population: FAS: Enrolled participants who have received at least one dose of treatment.
  The analysis for DOR assessed by investigator was based on the responders in the FAS of each cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 25 | 13
months | 5.8 [4.01 to 8.4] | 6.7 [4.2 to NA] — The upper limit is not calculable due to insufficient number of participants with events.

4. Secondary Outcome: Disease Control Rate (DCR), Assessed by ICR
Description: Disease control rate is defined as the percentage of participants who have a confirmed CR or PR or who have SD per RECIST 1.1, as assessed by ICR
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 77 | 40
Percentage | 72.7 [61.4 to 82.3] | 85 [70.2 to 94.3]

5. Secondary Outcome: Best Overall Response (BoR) , Assessed by ICR
Description: Best overall response is defined as participant's best confirmed response during their participation in the study, but prior to starting any subsequent anticancer therapy, up until RECIST 1.1-defined PD or the last evaluable assessment in the absence of RECIST 1.1-defined progression.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 77 | 40
Percentage
  Confirmed Partial Response | 33.8 | 45.0
  Confirmed Complete Response | 0 | 0

6. Secondary Outcome: Time To Response (TTR) , Assessed by ICR
Description: Time to response is defined as the time from the date of the first dose of study intervention until the date of first documented objective response, which is subsequently confirmed per RECIST 1.1
Time Frame: as for outcome 1
Population: RES: Enrolled participants who received at least one dose of study intervention and had measurable disease at baseline by ICR.
  The analysis for TTR assessed by ICR was based on the responders in the RES of each cohort.
Measure: Median (Inter-Quartile Range); unit: Month
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 26 | 18
Month | 1.5 [1.3 to 2.8] | 1.4 [1.3 to 2.7]

7. Secondary Outcome: Progression-Free Survival (PFS) , Assessed by ICR
Description: Progression-free survival is defined as time from the date of the first dose of study intervention until progression per RECIST 1.1, as assessed by ICR, or death due to any cause.
Time Frame: as for outcome 1
Population: FAS: Enrolled participants who have received at least one dose of treatment. Participants who were enrolled but did not subsequently receive study intervention are not included in the analysis.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 79 | 40
Month | 5.3 [4.2 to 6.9] | 7.4 [5.7 to NA] — The upper limit is not calculable due to insufficient number of participants with events.

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of the first dose of study intervention to the date of death due to any cause.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 79 | 40
Month | 13.5 [10.7 to NA] — The upper limit is not calculable. | NA [NA to NA] — The NAs are not calculable due to insufficient number of participants with events.

9. Secondary Outcome: Progression-Free Survival (PFS) , Assessed by Investigator
Description: Progression-free survival is defined as time from the date of the first dose of study intervention until progression per RECIST 1.1, as assessed by investigator, or death due to any cause.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 79 | 40
Month | 4.3 [4.0 to 5.6] | 7.0 [5.5 to 8.5]

10. Secondary Outcome: Disease Control Rate (DCR), Assessed by Investigator
Description: Duration of response is defined as the time from the date of first documented response (which is subsequently confirmed) until date of documented progression per RECIST 1.1, as assessed by investigator, or death due to any cause.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 77 | 40
Percentage | 76.6 [65.6 to 85.5] | 85.0 [70.2 to 94.3]

11. Secondary Outcome: Best Overall Response (BoR) , Assessed by Investigator
Description: as for outcome 5
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 77 | 40
Percentage
  Confirmed complete response | 0 | 0
  Confirmed partial response | 31.2 | 37.5

12. Secondary Outcome: Time To Response (TTR) , Assessed by Investigator
Description: as for outcome 6
Time Frame: as for outcome 1
Population: FAS: Enrolled participants who have received at least one dose of treatment. Participants who were enrolled but did not subsequently receive study intervention are not included in the analysis.
  The analysis for TTR assessed by investigator was based on the responders in the FAS of each cohort.
Measure: Median (Inter-Quartile Range); unit: Month
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 25 | 13
Month | 1.4 [1.4 to 1.6] | 1.4 [1.3 to 1.4]

13. Secondary Outcome: Pharmacokinetic Parameter: Area Under the Plasma Concentration- Time Curve (AUC) _ Total Anti-TROP2 Antibody
Description: PK parameters of Total Anti-TROP2 Antibody_Area under the curve
Time Frame: as for outcome 1
Population: PK analysis set:Enrolled participants who have received at least one dose of treatment and had measurable serum concentrations of Dato-DXd.
  The analysis for AUC was based on the patients with intensive PK collection of each cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 8 | 9
day*ug/mL | 713.9 (25.45) | 569.3 (24.47)

14. Secondary Outcome: Pharmacokinetic Parameter: Maximum Plasma Concentration (Cmax) _ Total Anti-TROP2 Antibody
Description: PK parameters of Total Anti-TROP2 Antibody_Maximum observed concentration
Time Frame: as for outcome 1
Population: PK analysis set:Enrolled participants who have received at least one dose of treatment and had measurable serum concentrations of Dato-DXd.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 79 | 40
ug/mL | 137.8 (19.09) | 121.1 (22.38)

15. Secondary Outcome: Pharmacokinetic Parameter: Area Under the Plasma Concentration- Time Curve (AUC) _Dato-DXd
Description: PK parameters of Dato-DXd_Area under the curve
Time Frame: as for outcome 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 8 | 9
day*ug/mL | 668.3 (21.11) | 504.5 (22.38)

16. Secondary Outcome: Pharmacokinetic Parameter: Maximum Plasma Concentration (Cmax) _ Dato-DXd
Description: PK parameters of Dato-DXd_Maximum observed concentration
Time Frame: as for outcome 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 79 | 40
ug/mL | 136.4 (20.18) | 115.4 (18.12)

17. Secondary Outcome: Pharmacokinetic Parameter: Area Under the Plasma Concentration- Time Curve (AUC) _ MAAA-1181a
Description: PK parameters of MAAA-1181a_Area under the curve
Time Frame: as for outcome 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 8 | 9
day*ng/mL | 17.60 (24.64) | 17.66 (33.09)

18. Secondary Outcome: Pharmacokinetic Parameter: Maximum Plasma Concentration (Cmax) _ MAAA-1181a
Description: PK parameters of MAAA-1181a_Maximum observed concentration
Time Frame: as for outcome 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 79 | 40
ng/mL | 2.484 (45.09) | 2.463 (42.31)

19. Secondary Outcome: Pharmacokinetic Parameter: Time to Maximum Plasma Concentration (Tmax) _Total Anti-TROP2 Antibody
Description: PK parameters of Total Anti-TROP2 Antibody_Time to maximum plasma concentration
Time Frame: as for outcome 1
Population: PK analysis set: Enrolled participants who have received at least one dose of treatment and had measurable serum concentrations of Dato-DXd.
Measure: Median (Full Range); unit: Hour
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 79 | 40
Hour | 2.00 [1.40 to 7.17] | 1.70 [0.90 to 6.83]

20. Secondary Outcome: Pharmacokinetic Parameter: Time to Maximum Plasma Concentration (Tmax) _Dato-DXd
Description: Time to maximum plasma concentration
Time Frame: as for outcome 1
Population: as for outcome 19
Measure: Median (Full Range); unit: h
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 79 | 40
h | 1.92 [1.12 to 7.17] | 1.77 [0.90 to 5.22]

21. Secondary Outcome: Pharmacokinetic Parameter: Time to Maximum Plasma Concentration (Tmax) _ MAAA-1181a
Description: PK parameters of MAAA-1181a_Time to maximum plasma concentration
Time Frame: as for outcome 1
Population: as for outcome 19
Measure: Median (Full Range); unit: Hour
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 79 | 40
Hour | 5.00 [1.67 to 24.22] | 4.98 [4.77 to 25.07]

22. Secondary Outcome: Immunogenicity of Dato-DXd
Description: The prevalence of ADA (positive at any visit)
Time Frame: as for outcome 1
Population: ADA Evaluable Set: Participants in the FAS with a non-missing baseline Dato-DXd ADA result and at least one post-baseline Dato-DXd ADA result.
Measure: Number; unit: percentage
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 75 | 38
percentage | 33.3 | 36.8

23. Secondary Outcome: Duration of Response (DoR), Assessed by ICR
Description: Duration of response is defined as the time from the date of first documented response (which is subsequently confirmed) until date of documented progression per RECIST 1.1, as assessed by ICR, or death due to any cause.
Time Frame: as for outcome 1
Population: RES: Enrolled participants who received at least one dose of study intervention and had measurable disease at baseline by ICR.
  The analysis for DOR assessed by ICR was based on the responders in the RES of each cohort.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | TNBC Cohort | NSCLC Cohort
Number analyzed (Participants) | 26 | 18
Month | 6.7 [4.53 to 12.6] | 8.3 [5.9 to NA] — The upper limit is not calculable due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: TNBC Cohort: Final analysis occurred 12 months after last participant of this cohort initiated Dato-DXd. NSCLC Cohort: Primary analysis occurred 6 months after last participant of this cohort initiated Dato-DXd.
Groups:
- Dato-DXd_TNBC; Dato-DXd_NSCLC: Description (Arm-group)
Arm/Group | Dato-DXd_TNBC | Dato-DXd_NSCLC
All-Cause Mortality (participants affected / at risk) | 43/79 | 9/40
Serious Adverse Events (participants affected / at risk) | 13/79 | 10/40
Other Adverse Events (participants affected / at risk) | 77/79 | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dato-DXd_TNBC (N=79) | Dato-DXd_NSCLC (N=40)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dato-DXd_TNBC (N=79) | Dato-DXd_NSCLC (N=40)
Constipation (Gastrointestinal disorders) | 19 (30) | 9 (11)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (4)
Mouth ulceration (Gastrointestinal disorders) | 8 (9) | 1 (3)
Nausea (Gastrointestinal disorders) | 34 (92) | 24 (81)
Stomatitis (Gastrointestinal disorders) | 38 (60) | 23 (39)
Vomiting (Gastrointestinal disorders) | 23 (51) | 13 (34)
Asthenia (General disorders) | 7 (16) | 9 (10)
Fatigue (General disorders) | 10 (11) | 5 (9)
Oedema peripheral (General disorders) | 4 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 20 (29) | 23 (34)
Covid-19 (Infections and infestations) | 8 (10) | 8 (9)
Conjunctivitis (Infections and infestations) | 1 (1) | 4 (4)
Suspected covid-19 (Infections and infestations) | 10 (11) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 10 (15) | 6 (8)
Leukopenia (Blood and lymphatic system disorders) | 10 (19) | 9 (16)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (12) | 2 (3)
Alanine aminotransferase increased (Investigations) | 21 (31) | 2 (3)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 (0) | 3 (3)
Amylase increased (Investigations) | 3 (4) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 21 (43) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 6 (8) | 4 (5)
Blood cholesterol increased (Investigations) | 4 (5) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 6 (7) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 12 (15) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 3 (3)
Lipase increased (Investigations) | 0 (0) | 3 (5)
Lymphocyte count decreased (Investigations) | 8 (16) | 2 (5)
Neutrophil count decreased (Investigations) | 26 (53) | 7 (9)
Platelet count decreased (Investigations) | 5 (7) | 3 (4)
Weight decreased (Investigations) | 10 (14) | 11 (12)
Weight increased (Investigations) | 4 (4) | 2 (2)
White blood cell count decreased (Investigations) | 25 (46) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 15 (23) | 10 (14)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 (13) | 3 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (15) | 3 (4)
Corneal epithelium defect (Eye disorders) | 4 (4) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 (6) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 11 (13) | 3 (6)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (9) | 4 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (12) | 7 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (8) | 2 (3)
Hypochloraemia (Metabolism and nutrition disorders) | 6 (9) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (23) | 7 (10)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (15) | 6 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 3 (8)
Dry eye (Eye disorders) | 4 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1)
Dizziness (Nervous system disorders) | 4 (9) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 4 (6) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Lacrimation increased (Eye disorders) | 1 (1) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (15) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 16 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 9 (11) | 4 (5)
Abdominal discomfort (Gastrointestinal disorders) | 5 (6) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-05-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT05460273/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT05460273/SAP_001.pdf